CLINICAL TRIAL: NCT01280214
Title: Peribulbar and Subconjunctival Kenalog Injection for Thyroid Orbitopathy
Brief Title: Local Triamcinolone Injection in Active Thyroid Orbitopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr Daniel Briscoe, Haemek Medical center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMC119710ctil
Record Dates: First submitted 2011-01-15; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Thyroid Disease
MeSH Terms: conditions — Thyroid Diseases | interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Triamcinolone (Experimental)
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone — Subconjunctival and peribulbar, 40 mg/ml, 3 monthly injection
  Other Names: kenalog

SUMMARY:
Comparing the effectiveness of subconjunctival and peribulbar Triamcinolone injection to systemic Steroid therapy for patients with active thyroid orbitopathy.

DETAILED DESCRIPTION:
Local Steroid treatment may help in active thyroid orbitopathy. till today, systemic Steroids are the treatment for active thyroid orbitopathy which is associated with systemic adverse effects.

In this study the investigators want to compare the effectiveness of local Triamcinolone therapy for active thyroid orbitopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Active thyroid orbitopathy according to clinical activity score>=3.

Exclusion Criteria:

* Intraorbital or active infections.
* Tuberculosis.
* Other orbital disease.
* Pregnancy.
* Compressive optic neuropathy.
* Systemic steroid therapy within 6 months of study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Comparing the effectiveness of subconjunctival and peribulbar Triamcinolone injection to systemic Steroid therapy for patients with active thyroid orbitopathy . | 6 months
  Every month, each participant will undergo several tests : blood sugar, full ocular examination, color test, visual field and ultrasound test for measuring the thickness of extraocular muscles.Clinical activity score for thyroid orbitopathy will be assesed too. The results of the clinical and ultrasonogrophic findings will determine the effectiveness of the treatment.
  A patient with deterioration of thyroid orbitopathy during the research, will be treated by systemic Steroids in addition to the local injections.

SECONDARY OUTCOMES:
To check if the level of TSH Receptor antibodies are affected by the local injection. | 4 months
  A blood test for TSH Receptor antibodies will be taken for every patient at the beginnig of the research and after 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Briscoe, MD, Study Chair — haemek medical center